CLINICAL TRIAL: NCT06533839
Title: Prevention of Parastomal Hernias With a Preformed Three-dimensional, Funnel-shaped Mesh. A Prospective, Multicenter and Randomized Study (PREVEMAC)
Brief Title: Prevention of Parastomal Hernias With a Preformed Three-dimensional, Funnel-shaped Mesh
Acronym: PREVEMAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/20
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia; end colostomy; prophylactic mesh

STUDY DESIGN:
Intervention Model Description: Multicentric randomised controlled trial
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPST mesh placement (Experimental): A three-dimensional, funnel-shaped mesh will be used.
  Interventions: Procedure: Permanent colostomy
- No mesh (Active Comparator): No mesh will be applied.
  Interventions: Procedure: Permanent colostomy

INTERVENTIONS:
Procedure: Permanent colostomy — A long-term (permanent) colostomy will be performed in the diseased colon or rectum.

SUMMARY:
Parastomal hernia (PH) remains a significant complication following stoma creation, boasting a considerable prevalence in the range of 30 to 50% within the first year post-surgery, a figure that climbs even higher when considering radiological evidence irrespective of clinical symptoms. A noteworthy one-third of these cases necessitate subsequent surgical interventions, yielding suboptimal outcomes both in the short and long term. The clinical manifestations of PH are diverse, ranging from mild inconveniences like fecal leakage and dermatitis to more severe and potentially life-threatening complications such as intestinal obstruction, hernia incarceration, and ischemia.

Various systematic reviews and meta-analyses have advocated for the adoption of prophylactic meshes, although defining precise incidence and recurrence rates has proven challenging due to methodological disparities across studies. Keyhole and modified Sugarbaker techniques dominate laparoscopic and robotic approaches, yet none offer ideal outcomes.

The aim of this study is to evaluate the decrease of postoperative parastomal hernia using this three-dimensional, funnel-shaped mesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a definitive colostomy confection
* Terminal colostomy confection
* ASA index III or inferior
* Patients who have given legat authorization to participate in the study

Exclusion Criteria:

* Lateral colostomy or a colostomy that will be removed posteriorly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative parastomal hernia prevention | up to one year post-intervention
  proportion of Postoperative parastomal hernias

SECONDARY OUTCOMES:
Postoperative parastomal hernia prevention | 5 years after surgery
  proportion of Postoperative parastomal hernias
readmissions for complications | up to one year post-intervention
  proportion of hospital readmissions
morbidity | up to one year post-intervention
  Comprehensive Complication Index (CCI) 20

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No